CLINICAL TRIAL: NCT02573051
Title: Misoprostol Plus Isosorbide Mononitrate Versus Misoprostol For Termination Of Anembryonic Pregnancy
Brief Title: Termination Of Anembryonic Pregnancy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANP
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Misoprostol; isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol plus isosorbide mononitrate (Active Comparator): this group will receive 800 µg of misoprostol (Misotac 200 µg Sigma for Pharmaceutical Industries) plus 40 mg isosorbide mononitrate (Effox 40 mg Minipharma Company) will be inserted into the posterior vaginal fornix
  Interventions: Drug: Misoprostol; Drug: Isosorbide mononitrate
- Misoprostol plus placebo (Active Comparator): This group will receive misoprostol 800 µg plus placebo in the same site.
  Interventions: Drug: Misoprostol; Other: placebo

INTERVENTIONS:
Drug: Misoprostol — 800 µg of misoprostol (Misotac 200 µg Sigma for Pharmaceutical Industries)
Drug: Isosorbide mononitrate — 40 mg isosorbide mononitrate (Effox 40 mg Minipharma Company)
  Arms: Misoprostol plus isosorbide mononitrate
Other: placebo
  Arms: Misoprostol plus placebo

SUMMARY:
Anembryonic pregnancy is a leading cause of early miscarriage. The American Pregnancy Association estimates that blighted ovum causes approximately 50 percent of all first-trimester miscarriages. About 20 percent of all pregnancies result in miscarriage.

In general, there are 3 options for management of anembryonic pregnancy: expectant, medical, and surgical management. Expectant management consists of no intervention and awaiting natural passage of tissue. Medical management uses medication to expel uterine tissue. Surgical management is defined by mechanical removal of tissue from the uterus.

Medical management allows patients to avoid surgery and anesthesia. Patients may also feel that medical management is more private, and under their control. Several medications have been studied for medical management.

Misoprostol, a prostaglandin E1 analogue, is a uterotonic that results in cervical softening and contractions that expel the products of conception. It may be administered vaginally, orally, buccally, or sublingually. Adverse effects vary based on route of administration.

There is published literature on a wide range of therapeutic misoprostol regimens. Optimal dose and route of administration of misoprostol have not been determined by randomized trials. Overall, misoprostol is safe and well-tolerated.

Patients receiving misoprostol vaginally rather than orally have decreased adverse gastrointestinal effects and prolonged duration of action.

Oral misoprostol is less effective than vaginal misoprostol in emptying the uterus. Sublingual misoprostol is equivalent to vaginal misoprostol in inducing complete uterine emptying but is associated with more frequent diarrhea.

When compared with lower dosages, a dose of 800 µg vaginal misoprostol is more effective at completing uterine emptying, although it results in a similar incidence of nausea. Based on international trials in settings with limited resources, WHO recommends a single vaginal dose of 800 µg misoprostol for medical management of anembryonic pregnancy. Routes of misoprostol administration include oral, vaginal, buccal or rectal. Vaginal misoprostol is associated with a greater overall exposure to the drug and greater effects on the cervix and uterus.

Isosorbide mononitrate (IMN) is a drug used principally in the treatment of angina pectoris, which acts by dilating the blood vessels so as to reduce blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥20years old.
* No vaginal bleeding.
* No dilation of internal os.
* Gestational age: from 8-11weeks.
* Gestational sac with a mean gestational sac diameter (MGD) greater than 25 mm and no yolk sac, or an MGD >25 mm with no embryo.

Exclusion Criteria:

* Patients with excessive vaginal bleeding (soaking more than a pad per day).
* Patients with dilated cervix.
* Patients with allergy either to misoprostol or isosorbide mononitrate.
* Those who will be insisted on D and C will be excluded from the study.
* Women will be excluded from the study if they are anemic (hemoglobin less than 11 g/dl).
* Hemo-dynamically unstable with signs of pelvic infection and/or sepsis.
* Suffering from a clotting disorder or using anticoagulants.
* Women with uterine pathology such as myomas or malformation.
* Women had previous caesarian section.
* Asthmatic patients.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
The measurement of endometrial thickness by ultrasound in mm | 6 months
  Complete expulsion of remnant of conception is considered if endometrial thickness less than 10 mm and if more than 10 mm it considered incomplete expulsion.

SECONDARY OUTCOMES:
Induction - abortion interval in hours | 6 months
  The period from the start of administration of misoprostol until complete abortion
Induction dilatation interval in hours | 6 month
  The period from the start of administration of misoprostol until the start of cervical dilatation measured during per vagina (P/V) examination
The occurrence of sever uncontrolled lower abdominal pain by visual analogue scale | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt